CLINICAL TRIAL: NCT06898957
Title: A Phase 1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Tarlatamab in Combination With YL201 With or Without Anti-PD-L1 in Subjects With Extensive Stage Small Cell Lung Cancer
Brief Title: Study of Tarlatamab in Combination With YL201 With or Without Anti-programmed Death Ligand 1 (PD-L1) in Participants With Extensive Stage (ES) Small Cell Lung Cancer (SCLC)
Acronym: (DeLLphi-310)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: MediLink (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20240124
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Cancer
Keywords: Small cell lung cancer; SCLC; Tarlatamab; YL201; Anti-PD-L1; Atezolizumab; Durvalumab
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Exploration (Part 1) (Experimental): Multiple dose levels of YL201 will be explored in combination with tarlatamab administered intravenously (IV) at a fixed dose using one-step dosing.
  Interventions: Drug: YL201; Drug: Tarlatamab
- Dose Expansion (Part 2) (Experimental): YL201 will be administered at the selected maximum tolerated combination dose (MTCD) or recommended phase 2 dose (RP2D) in combination with tarlatamab administered IV at a fixed dose.
  Interventions: Drug: YL201; Drug: Tarlatamab
- Triplet Combination (Part 3) (Experimental): YL201 will be administered at MTCD or RP2D in combination with tarlatamab and an anti-PD-L1 (atezolizumab or durvalumab) administered IV at a fixed dose.
  Interventions: Drug: YL201; Drug: Tarlatamab; Drug: Atezolizumab; Drug: Durvalumab

INTERVENTIONS:
Drug: YL201 — YL201 will be administered as an IV infusion.
Drug: Tarlatamab — Tarlatamab will be administered as an IV infusion.
Drug: Atezolizumab — Atezolizumab will be administered as an IV infusion.
  Arms: Triplet Combination (Part 3)
Drug: Durvalumab — Durvalumab will be administered as an IV infusion.
  Arms: Triplet Combination (Part 3)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of tarlatamab in combination with YL201 with or without anti-PD-L1.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥ 18 years of age (or legal adult age within country) at time of signing informed consent.
* Participants with histologically or cytologically confirmed ES-SCLC.
* For Parts 1 and 2, participant must have ES-SCLC that has progressed or recurred following at least 1 line of platinum-based anti-cancer therapy.
* For Part 3, participants must have ES-SCLC and no prior systemic treatment for ES SCLC other than 1 cycle of platinum-based chemotherapy, etoposide, and PD-(L)1 inhibitor in the first-line setting.
* At least 1 measurable lesion as defined by RECIST 1.1.
* Participants must have adequate organ function (cardiac, pulmonary, kidney, bone marrow, and liver).

Exclusion Criteria:

* Prior delta-like ligand 3 (DLL3) or B7 homolog 3 (B7-H3) targeted therapy.
* Prior exposure to topoisomerase I inhibitors or antibody-drug conjugate (ADC) with topoisomerase I inhibitor payload.
* Symptomatic central nervous system (CNS) metastases. Note: Participants with asymptomatic brain metastases are eligible as defined in the protocol.
* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required corticosteroids, current ILD/pneumonitis, or suspected ILD/pneumonitis that cannot be ruled out by imaging at screening.
* Baseline requirement of supplemental oxygen.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2031-04-23 (Estimated); Study Completion 2031-04-23 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting toxicities (DLTs) | Up to Day 21
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to 3.5 Years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 3.5 Years
Duration of Response (DOR) per RECIST 1.1 | Up to 3.5 Years
Time to Response (TTR) per RECIST 1.1 | Up to 3.5 Years
Disease Control Rate (DCR) per RECIST 1.1 | Up to 3.5 Years
Progression-free Survival (PFS) per RECIST 1.1 | Up to 3.5 Years
Time to Progression (TTP) per RECIST 1.1 | Up to 3.5 Years
Time to Subsequent Therapy | Up to 3.5 Years
Overall Survival (OS) | Up to 3.5 Years
Maximum Serum Concentration (Cmax) of Tarlatamab | Up to Week 36
Minimum Serum Concentration (Cmin) of Tarlatamab | Up to Week 36
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval for Tarlatamab | Up to Week 36
Half-life (t1/2) of Tarlatamab | Up to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (36):
- United States (11):
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Siteman Cancer Center, St Louis, Missouri
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Sanford Oncology Clinic and Pharmacy, Sioux Falls, South Dakota
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- CHU de Quebec Hopital de l Enfant Jesus, Québec, Quebec, Canada
- China (3):
  - Shandong Cancer Hospital, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Fujian Cancer Hospital, Fuzhou
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Universitaetsklinikum Essen, Essen, Germany
- Greece (4):
  - Henry Dunant Hospital Center, Athens
  - Alexandra Hospital, Athens
  - European Interbalkan Medical Center, Thessaloniki
  - Iatriko Diavalkaniko Thessalonikis, Thessaloniki
- Hungary (2):
  - Semmelweis Egyetem, Budapest
  - Clinexpert Kft Bugat Pal Korhaz, Gyöngyös
- Italy (3):
  - Istituto di Candiolo Fondazione del Piemonte per l Oncologia IRCCS, Candiolo to
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola (FC)
  - Azienda Socio Sanitaria Territoriale Grande Ospedale Metropolitano Niguarda, Milan
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Universitari Vall d Hebron, Barcelona, Catalonia
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request .De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com